CLINICAL TRIAL: NCT04583319
Title: A Prospective, Non-interventional Study for Validation of a Rapid, Non-invasive IVD as a Point-of-care Test for Diagnosis of SARS-COV-2 Infection
Brief Title: Validation of a Rapid, Non-invasive Point-of-care IVD Test for Diagnosis of SARS-COV-2 (COVID-19) Infection
Acronym: EasyCov
Status: Completed | Type: Observational
Sponsor: Firalis SA (Industry)
Collaborators: Istanbul University (Other)
Responsible Party: Sponsor
Other Study IDs: ST0194
Record Dates: First submitted 2020-09-30; First posted 2020-10-12 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: SARS-CoV
Keywords: SARS Coronavirus; Coronavirus; Covid-19
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples of Subjects will be collected in a FDA approved collection device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SARS-CoV-2 Positive: patients tested positive for SARS-CoV-2 by routine Turkish MOH and FDA approved RT-PCR IVD test.
  Interventions: Diagnostic Test: EasyCov POC
- SARS-CoV-2 Negative: participants tested negative for SARS-CoV-2 by routine Turkish MOH and FDA approved RT-PCR IVD test.
  Interventions: Diagnostic Test: EasyCov POC

INTERVENTIONS:
Diagnostic Test: EasyCov POC — Saliva samples will be collected according to the sampling protocol defined each for EASYCOV test. The EasyCoV test will be performed at the beginning of the study before obtaining the routine RT- PCR test results. The operators performing this test will be blinded from the routine RT-PCR results.

SUMMARY:
A prospective non-interventional study to evaluate the performance of EASYCOV IVD as point-of-care (POC) test by comparing SARS-CoV-2 positive patients with SARS-CoV-2 negative controls on paired specimens (nasopharyngeal swabs & saliva samples).

DETAILED DESCRIPTION:
A prospective non-interventional study to evaluate the performance of EASYCOV IVD as point-of-care (POC) test by comparing SARS-CoV-2 positive patients with SARS-CoV-2 negative controls on paired specimens (nasopharyngeal swabs & saliva samples).

The operators performing the diagnostic tests will be blinded from the RT-PCR results (i.e. participant's group will be anonymized). Participants who have been tested by an routineTurkish MOH and FDA EUA approved RT-PCR test using nasopharyngeal swabs will be included in the study to perform the EASYCOV IVD tests in a POC setting.

Primary Objective:

• To evaluate the performance of EasyCov IVD as a point-of-care (POC) test performed on saliva samples for the diagnosis of SARS-CoV-2 infection by comparing it to a Turkish MOH and FDA EUA approved RT-PCR test performed on nasopharyngeal samples.

Secondary Objectives:

• Collection and storage of saliva samples, nasopharyngeal swabs at D0 to perform future COVID-19 related research projects and validation of future generations of EASYCOV assays as well as exploratory studies to find candidate biomarkers for Covid-19.

160 participants will be included in 1:1 ratio: 80 SARS-CoV-2 positive and 80 SARS-CoV-2 negative by a Turkish MOH and FDA approved RT-PCR IVD test

ELIGIBILITY:
Inclusion Criteria:

Non-specific inclusion criteria:

1. Participant aged 18 and above
2. Participant agreeing to follow the study procedures
3. Participant able to understand the purpose, nature and methodology of the study
4. Participant having signed the informed consent

Specific inclusion criteria:

SARS-COV-2 positive patients - Participants tested positive for the SARS-COV-2 by the routine Turkish MOH and FDA approved RT-PCR method.

SARS-COV-2 negative controls

- Participants tested negative for the SARS-COV-2 by the routine Turkish MOH and FDA approved RT-PCR method.

Exclusion Criteria:

* Minors, persons deprived of their liberty, protected adults or vulnerable persons.
* Refusal to sign the consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment will be carried out on patients suspected to have contracted COVID-19 and to be screened by RT-PCR test, according to decision of her/his physician. These patients are routinely screened by a Turkish MOH and FDA approved RT-PCR test for COVID-19 and will be allocated to SARS-COV-2 Positive or Control group based on results obtained from RT-PCR.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Positive percent agreement (PPA) | 1 month
  A positive percent agreement (PPA) of EASYCOV PoC assay will be corroborated with the routine Turkish MOH and FDA approved reference method RT-PCR using nasopharyngeal samples.

SECONDARY OUTCOMES:
Performance | 1 month
  The performance (accuracy, sensitivity, specificity, positive predictive value, negative predictive value) of EASYCOV POC assay will be evaluated compared to the routine Turkish MOH and FDA approved RT-PCR method using nasopharyngeal samples.

CONTACTS AND LOCATIONS:
Overall Officials: Arif Atahan, Prof.MD, Principal Investigator — Istanbul University Istanbul Faculty of Medicine (ITF), Turkey
Locations (1):
- Istanbul University Istanbul Faculty of Medicine (ITF), Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No